CLINICAL TRIAL: NCT05209256
Title: Alflutinib Versus Alflutinib Plus Chemotherapy for Nonesmall Cell Lung Cancer With EGFR (T790M)- Associated Resistance to Initial EGFR Inhibitor Treatment: An Open-label, Randomised Phase 2 Clinical Trial
Brief Title: Alflutinib Versus Alflutinib Plus Chemotherapy for NSCLC
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: The First Affiliated Hospital of Henan University of Science and Technology (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ALF-IN-NSCLC-001
Record Dates: First submitted 2022-01-09; First posted 2022-01-26 (Actual); Last update posted 2022-01-26 (Actual); Status verified 2021-10

CONDITIONS: NSCLC
Keywords: NSCLC ，EGFR(T790M)，alflutinib
MeSH Terms: interventions — Drug Therapy; Pemetrexed; aflutinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Alflutinib plus chemotherapy (Experimental): Those in the combination group received concurrent alflutinib (80 mg daily), as well as carboplatin (area under the curve [AUC] of 5 on day 1) and pemetrexed (500 mg/m2 on day 1) in a 3-week cycle for up to four cycles, followed by maintenance on alflutinib and pemetrexed until disease progression, unacceptable toxicity, or death.
  Interventions: Drug: Alflutinib plus chemotherapy
- chemotherapy (Sham Comparator): arboplatin (area under the curve [AUC] of 5 on day 1) and pemetrexed (500 mg/m2 on day 1) in a 3-week cycle for up to four cycles, followed by maintenance on alflutinib and pemetrexed until disease progression, unacceptable toxicity, or death.
  Interventions: Drug: Chemotherapy

INTERVENTIONS:
Drug: Chemotherapy — Patients in the alflutinib group received alflutinib (80 mg daily) until disease progression, unacceptable toxicity, or death.
  Other Names: pemetrexed; Pulaile
  Arms: chemotherapy
Drug: Alflutinib plus chemotherapy — Those in the combination group received concurrent alflutinib (80 mg daily), as well as carboplatin (area under the curve [AUC] of 5 on day 1) and pemetrexed (500 mg/m2 on day 1) in a 3-week cycle for up to four cycles, followed by maintenance on alflutinib and pemetrexed until disease progression, unacceptable toxicity, or death.
  Other Names: AST2818; Pulaile
  Arms: Alflutinib plus chemotherapy

SUMMARY:
Aim: the aim of this study is to investigated whether the combination of alflutinib with cytotoxic chemotherapy might hold additive efficacy, as well as tolerability .

DETAILED DESCRIPTION:
alflutinib is a third-generation epidermal growth factor receptor (EGFR) tyrosine kinase inhibitor (TKI) that is active in the central nervous system (CNS) and which potently and selectively inhibits mutant forms of EGFR with both TKI-sensitising (activating) mutations and the T790M resistance-conferring mutation. However, resistance to alflutinib inevitably emerges. One promising strategy to further improve patient prognosis and to approach a cure is combination therapy with alflutinib and other agents such as cytotoxic chemotherapeutic drugs.

ELIGIBILITY:
Inclusion Criteria:

* histologically or cytologically diagnosed non-squamous NSCLC of stage IIIB or IV (based on the 7th edition of the TNM classification) or recurrent;
* an EGFR mutation, including an exon-19 deletion (Ex19del), L858R, or other (L861Q, G719A, G719C, or G719S), as well as the T790M mutation of EGFR as detected in a tissue or liquid biopsy sample obtained after disease progression during first-line EGFR-TKI (gefitinib, erlotinib, or afatinib) treatment;
* WHO performance status of 0 or 1;
* no prior neoadjuvant or adjuvant chemotherapy in the 12 months preceding study enrollment;
* adequate bone marrow reserve and organ function.

Exclusion Criteria:

* treatment with an EGFR-TKI within 7 days of the first dose of the study treatment;
* symptomatic CNS metastases;
* evidence of interstitial pneumonia, pulmonary fibrosis, or radiation pneumonitis requiring steroid treatment as revealed by a computed tomography (CT) scan.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2022-03-01 (Estimated); Primary Completion 2024-01 (Estimated); Study Completion 2025-01 (Estimated)

PRIMARY OUTCOMES:
PFS | 16 weeks
  Disease-free survival

SECONDARY OUTCOMES:
Objective remission rate (ORR) | 16 weeks
  Objective remission rate
Disease Control Rate ( DCR) | 16 weeks
  Disease Control Rate

CONTACTS AND LOCATIONS:
Overall Officials: Xinshuai Wang, PHD, Principal Investigator — The First Affiliated Hospital of Clinical Medicine of Henan University of Science and Technology; Guoqiang Kong, MD, Principal Investigator — The First Affiliated Hospital of Clinical Medicine of Henan University of Science and Technology; Xiaozhi Yuan, MD, Principal Investigator — The First Affiliated Hospital of Clinical Medicine of Henan University of Science and Technology; Jing Ren, MD, Principal Investigator — The First Affiliated Hospital of Clinical Medicine of Henan University of Science and Technology

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Garcia-Campelo R, Arrieta O, Massuti B, Rodriguez-Abreu D, Granados ALO, Majem M, Vicente D, Lianes P, Bosch-Barrera J, Insa A, Domine M, Reguart N, Guirado M, Sala MA, Vazquez-Estevez S, Caro RB, Drozdowskyj A, Verdu A, Karachaliou N, Molina-Vila MA, Rosell R; Spanish Lung Cancer Group (SLCG). Combination of gefitinib and olaparib versus gefitinib alone in EGFR mutant non-small-cell lung cancer (NSCLC): A multicenter, randomized phase II study (GOAL). Lung Cancer. 2020 Dec;150:62-69. doi: 10.1016/j.lungcan.2020.09.018. Epub 2020 Oct 3. PMID 33070053
- [Background] Griesinger F, Eberhardt W, Nusch A, Reiser M, Zahn MO, Maintz C, Bernhardt C, Losem C, Stenzinger A, Heukamp LC, Buttner R, Marschner N, Janicke M, Fleitz A, Spring L, Sahlmann J, Karatas A, Hipper A, Weichert W, Heilmann M, Sadjadian P, Gleiber W, Grah C, Waller CF, Reck M, Rittmeyer A, Christopoulos P, Sebastian M, Thomas M; CRISP Registry Group. Biomarker testing in non-small cell lung cancer in routine care: Analysis of the first 3,717 patients in the German prospective, observational, nation-wide CRISP Registry (AIO-TRK-0315). Lung Cancer. 2021 Feb;152:174-184. doi: 10.1016/j.lungcan.2020.10.012. Epub 2020 Nov 2. PMID 33358484
- [Background] Hochmair MJ, Morabito A, Hao D, Yang CT, Soo RA, Yang JC, Gucalp R, Halmos B, Marten A, Cufer T. Sequential afatinib and osimertinib in patients with EGFR mutation-positive non-small-cell lung cancer: final analysis of the GioTag study. Future Oncol. 2020 Dec;16(34):2799-2808. doi: 10.2217/fon-2020-0740. Epub 2020 Aug 28. PMID 32854536
- [Background] Imyanitov EN, Iyevleva AG, Levchenko EV. Molecular testing and targeted therapy for non-small cell lung cancer: Current status and perspectives. Crit Rev Oncol Hematol. 2021 Jan;157:103194. doi: 10.1016/j.critrevonc.2020.103194. Epub 2020 Dec 11. PMID 33316418
- [Background] Kayatani H, Ohashi K, Ninomiya K, Makimoto G, Nishii K, Higo H, Watanabe H, Kano H, Kato Y, Ninomiya T, Kubo T, Rai K, Ichihara E, Hotta K, Tabata M, Maeda Y, Kiura K. Beneficial effect of erlotinib and trastuzumab emtansine combination in lung tumors harboring EGFR mutations. Biochem Biophys Res Commun. 2020 Nov 12;532(3):341-346. doi: 10.1016/j.bbrc.2020.07.055. Epub 2020 Sep 2. PMID 32888648
- [Background] Mok TS, Cheng Y, Zhou X, Lee KH, Nakagawa K, Niho S, Chawla A, Rosell R, Corral J, Migliorino MR, Pluzanski A, Noonan K, Tang Y, Pastel M, Wilner KD, Wu YL. Updated Overall Survival in a Randomized Study Comparing Dacomitinib with Gefitinib as First-Line Treatment in Patients with Advanced Non-Small-Cell Lung Cancer and EGFR-Activating Mutations. Drugs. 2021 Feb;81(2):257-266. doi: 10.1007/s40265-020-01441-6. PMID 33331989
- [Background] Nakahara Y, Matsutani T, Igarashi Y, Matsuo N, Himuro H, Saito H, Yamada K, Murotani K, Hoshino T, Azuma K, Sasada T. Clinical significance of peripheral TCR and BCR repertoire diversity in EGFR/ALK wild-type NSCLC treated with anti-PD-1 antibody. Cancer Immunol Immunother. 2021 Oct;70(10):2881-2892. doi: 10.1007/s00262-021-02900-z. Epub 2021 Mar 9. PMID 33751180
- [Background] Nakashima K, Ozawa Y, Daga H, Imai H, Tamiya M, Tokito T, Kawamura T, Akamatsu H, Tsuboguchi Y, Takahashi T, Yamamoto N, Mori K, Murakami H. Osimertinib for patients with poor performance status and EGFR T790M mutation-positive advanced non-small cell lung cancer: a phase II clinical trial. Invest New Drugs. 2020 Dec;38(6):1854-1861. doi: 10.1007/s10637-020-00943-0. Epub 2020 May 18. PMID 32424780